CLINICAL TRIAL: NCT02515110
Title: Hypofractionated Regional Nodal Irradiation Phase 2 Clinical Trial for Women With Breast Cancer - HeNRIetta
Brief Title: Hypofractionated Regional Nodal Irradiation Clinical Trial for Women With Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15-10994; HM20004979 (Other: IRB); NCI-2015-01317 (Registry Identifier: CTRP)
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Node-positive Breast Cancer; Breast Adenocarcinoma; Invasive Breast Carcinoma; Lobular Breast Carcinoma In Situ
Keywords: lumpectomy; mastectomy without reconstruction; mastectomy with reconstruction; Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; HER2/Neu Positive; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (EBRT) (Experimental): External Beam Radiation Therapy (EBRT). Within 10 weeks after the last breast cancer surgery or the last dose of adjuvant chemotherapy, patients undergo hypofractionated RNI five days a week over 3-4 weeks.
  The two subgroups are Cohort (A) sentinel lymph node (SLN) and Cohort (B) axillary lymph node (ALN) dissection. They are categorized depending on type of axillary surgery and treatment group. The type of axillary surgery is Sentinel lymph node (SLN) biopsy only vs axillary dissection with or without previous SLN biopsy. The treatment groups are lumpectomy vs mastectomy vs mastectomy/reconstruction.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo hypofractionated RNI
  Other Names: Definitive Radiation Therapy; EBRT; External Beam RT; RNI
Other: Questionnaire Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
Single-arm, phase 2 study evaluating hypofractionated irradiation of breast and regional nodes in women with breast cancer. Patients will be grouped in 3 surgery-related treatment groups: 1) An intact breast following lumpectomy; 2) plans for loco regional external beam radiotherapy (EBRT) following mastectomy (with or without plans for reconstruction); and 3) plans for locoregional EBRT following mastectomy with reconstruction.

Patients will be assessed for lymphedema, arm function, breast or chestwall pain, other EBRT-related adverse events, and, for patients who had a lumpectomy or mastectomy with reconstruction, cosmetic outcome.

DETAILED DESCRIPTION:
The HeNRIetta Trial is a phase 2 non-randomized clinical trial to evaluate the safety and effectiveness of hypofractionated RNI for women with resected node-positive breast cancer. The study hypothesis is that a 3-4 week hypofractionated course of post-lumpectomy or postmastectomy EBRT is as safe and effective as the biologically equivalent dose given in conventional fractionation over 5-7 weeks.

Eligible patients are women ≥ 40 years old who have undergone definitive surgery for node-positive breast cancer. Surgery may have been lumpectomy, mastectomy without reconstruction, or mastectomy with reconstruction. Nodal staging may have been performed by only sentinel lymph node (SLN) or by axillary lymph node (ALN) dissection. Patients may have received neoadjuvant or adjuvant chemotherapy at the discretion of the treating medical oncologist.

Breast and RNI will be administered to 42.56 Gy in 16 fractions. (RNI will exclude the axilla in patients who have had an ALN dissection.) A treatment boost of 4 to 6 fractions of 2.66 Gy/fraction to the lumpectomy cavity will be included for all patients who have had lumpectomy; a chestwall boost (4 to 6 fractions of 2.66 Gy/fraction) will be administered to patients who had mastectomy (with or without reconstruction) and close (< 2 mm) surgical margins. Total number of EBRT fractions will be 20 to 22 with a boost; 16 without a boost.

Bilateral measurements of arm circumference will be used to assess lymphedema by comparing the ipsilateral arm to the contralateral arm. Patients will also be assessed for and will complete questionnaires related to lymphedema, decreased arm function, breast and chestwall pain, other EBRT-related toxicities, cosmetic outcome, and local, regional, and distant breast cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of 70-100%
* Histologic documentation of invasive adenocarcinoma of the breast
* One of the breast disease stages listed below:

  * Note: In the definitions below, definitive surgery is defined as the final surgery performed to obtain clear surgical margins
  * Neoadjuvant chemotherapy was not administered ** If neoadjuvant chemotherapy was NOT administered, pathologic staging must be T1-3, N1-2a following definitive surgery
  * Neoadjuvant chemotherapy was administered

    * If prior to initiation of neoadjuvant chemotherapy clinical staging was T1-3, N0, pathologic staging must be T1-3, N1-2a following definitive surgery
    * If prior to initiation of neoadjuvant chemotherapy clinical staging was T1-3, N1, pathologic staging must be T0-3, N0-2a following definitive surgery
    * If prior to initiation of neoadjuvant chemotherapy there was cytologic or pathologic confirmation of axillary nodal involvement (per any of the criteria listed below), pathologic staging must be T0-3, N0-2a following definitive surgery

      * Positive fine-needle aspiration (FNA) (ie, demonstrating malignant cells)
      * Positive core needle biopsy (ie, demonstrating invasive adenocarcinoma)
      * Positive sentinel lymph node biopsy (ie, demonstrating invasive adenocarcinoma)
* Complete resection of known breast disease by one of the following surgeries:

  * Lumpectomy with sentinel lymph node or axillary lymph node dissection
  * Mastectomy alone with sentinel lymph node or axillary lymph node dissection
  * Mastectomy plus reconstruction with sentinel lymph node or axillary lymph node dissection
* Margins of the resected specimen or re-excision specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the pathologist

  * Notes: Additional operative procedures may be performed to obtain clear margins; focally positive margins are acceptable based on technical feasibility of additional surgery and/or the potential for benefit with further surgery based on the extent and location of the positive margin (eg, focally positive deep margin at the pectoralis fascia); also, patients with margins positive for lobular carcinoma in situ (LCIS) are eligible without additional resection
* Estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2) testing performed on the primary breast tumor; when applicable, testing must have been performed prior to neoadjuvant chemotherapy
* Interval between the last surgery for breast cancer (including re-excision of margins) or the completion of adjuvant chemotherapy and study enrollment must be =< 56 days (ie, a maximum of 8 weeks)

  * Note: Radiotherapy must begin within 10 weeks following the last surgery for breast cancer or the last dose of adjuvant chemotherapy
* Recovery from surgery with the incision completely healed and no signs of infection
* If adjuvant chemotherapy was administered, chemotherapy-related toxicity that may interfere with delivery of external beam radiation therapy (EBRT) should have resolved
* Women who are not postmenopausal or have not undergone hysterectomy must have a documented negative pregnancy test within 14 days prior to study registration

  * Note: Postmenopausal is defined as one or more of the following:
  * Age >= 60 years
  * Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
  * Bilateral oophorectomy
* Women of child-bearing potential (WCBP) must agree to use a medically accepted form of pregnancy prevention for the duration of study treatment
* Ability to understand and willingness to sign the consent form written in English pregnancy test within 14 days prior to study registration

  * Note: Postmenopausal is defined as one or more of the following:
  * Age >= 60 years
  * Age < 60 years and amenorrheic for at least 1 year with follicle-stimulating hormone (FSH) and plasma estradiol levels in the postmenopausal range
  * Bilateral oophorectomy
* Women of child-bearing potential (WCBP) must agree to use a medically accepted form of pregnancy prevention for the duration of study treatment
* Ability to understand and willingness to sign the consent form written in English

Exclusion Criteria:

* Known definitive clinical or radiologic evidence of metastatic disease
* T4 tumors including inflammatory breast cancer
* Clinical nodal staging of N2 or N3 disease
* Pathologic nodal staging of N2b, N2c, or N3 disease
* Microscopic positive margins after definitive surgery

  * Note: Patients with microscopically focally positive margins following lumpectomy or mastectomy are not excluded if re-excision is not technically feasible and/or there is no benefit to further surgery based on the extent and location of the positive margin
* Any history, not including the index cancer, of ipsilateral or contralateral invasive breast cancer or ipsilateral or contralateral DCIS treated with radiation therapy (RT)

  * Note: Patients with synchronous or previous ipsilateral LCIS are eligible
* Any radiation therapy (RT) for the currently diagnosed breast cancer prior to study enrollment
* History of ipsilateral or contralateral breast or thoracic RT for any condition
* History of ipsilateral or contralateral axillary surgery for any condition
* History of lymphedema involving the ipsilateral or contralateral arm at present or at any time in the past
* Synchronous contralateral breast cancer requiring RT
* Overall geometry (eg, breast size if intact breast) precludes the ability to achieve dosimetric requirements

  * Note: Set-up devices for breast positioning are permitted
* Unresolved post-surgical complications (eg, significant infection) with healing difficulties
* Active collagen vascular disease, specifically dermatomyositis with a creatine phosphokinase (CPK) level above normal or with an active skin rash, systemic lupus erythematosus, or scleroderma
* Pregnancy or breastfeeding
* Diagnosis or treatment for a non-breast malignancy within 5 years of study registration, with the following exceptions: complete resection of basal cell carcinoma or squamous cell carcinoma of the skin and any in situ malignancy after curative therapy
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2015-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the cumulative incidence of lymphedema during the 3 years following completion of hypofractionated radiation treatment | 3 years
  Incidence of lymphedema defined as ≥ 10% increase in arm circumference over baseline circumference compared to the contralateral arm measured every 6 months from the time of initiation of hypofractionated irradiation of breast and regional nodes through 3 years following the completion of radiation therapy in 2 patient cohorts:
  * Patients who have only had SLN biopsy for axillary staging
  * Patients who have had ALN dissection for axillary staging

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Arthur, M.D., Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Healthcenter, South Hill, Virginia